CLINICAL TRIAL: NCT04453579
Title: Was it Right to Stop Bariatric Surgery During COVID-19 Lockdown?
Brief Title: Bariatric Surgery During Lockdown, Impact of COVID-19 on Physical and Mental Health
Status: Completed | Type: Observational
Sponsor: University of Rome Tor Vergata (Other)
Responsible Party: Principal Investigator, Paolo Gentileschi, Head of Bariatric Unit, University of Rome Tor Vergata
Other Study IDs: UNRomeB
Record Dates: First submitted 2020-06-29; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Obese; Morbid Obesity
Keywords: Bariatric surgery; Covid-19; Obesity; Mental health; Eating disorder
MeSH Terms: conditions — Obesity; Obesity, Morbid; COVID-19; Psychological Well-Being; Feeding and Eating Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 116 patients completed a survey: 116 patients were assessed during the Italian lockdown by means of a telephone interview performed by a trained researcher. The interview was composed of socio-demographic items (e.g. employed before and during the lockdown, own accommodation during lockdown etc.) and questions about physical and mental health in relation to the COVID-19 emergency
  Interventions: Behavioral: Telephonic interview during the Italian lockdown.

INTERVENTIONS:
Behavioral: Telephonic interview during the Italian lockdown. — The interview was composed of socio-demographic items lockdown, and dichotomous questions about physical and mental health in relation to the COVID-19 emergency

SUMMARY:
From the beginning of March 2020, lockdown regimens prevented patients with obesity from receiving bariatric surgery. Surgical emergencies and oncological procedures were the only operations allowed in public hospitals. Consequently, patients with morbid obesity were put in a stand-by situation. With the aim at exploring physical and psychological conditions of the investigators future bariatric surgery patients, the investigators built a Questionnaire concerning obesity and COVID-19.

DETAILED DESCRIPTION:
Introduction: the investigators present an investigation about the impact of COVID-19 on individuals suffering from severe obesity that were in the waiting list for bariatric surgery. Worldwide and in Italy bariatric procedures are considered as elective surgery and therefore were interrupted during the lockdown. The patients are well-known victim of stigma, social discrimination and the majority of them is affected by maladaptive eating behaviors that are supposed to worsen due to the isolation, absence of healthcare check-up and alarming pandemic scenario.the investigators performed telephonic interview providing an ad hoc questionnaire with the aim to explore their emotional and physical status.

Method: A total of 116 bariatric surgery candidates were approached using a telephonic interview during the Italian lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Severe Obesity with BMI > 35 kg/m2

Exclusion Criteria:

* Alcoholism
* Drug addiction

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From March 9th to May 4th 2020, 116 bariatric surgery candidates were approached using a telephonic interview during the Italian lockdown. The interview was composed of socio-demographic items and dichotomous about physical and mental health in relation to the COVID-19 emergency.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Psychological conditions | 2 months
  exploring physical and psychological conditions of our future bariatric surgery patients

CONTACTS AND LOCATIONS:
Overall Officials: paolo gentileschi, MD, Principal Investigator — University Hospital of Tor Vergata, Rome, Italy
Locations (1):
- Michela Campanelli, Rome, RM, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Epidemiology Working Group for NCIP Epidemic Response, Chinese Center for Disease Control and Prevention. [The epidemiological characteristics of an outbreak of 2019 novel coronavirus diseases (COVID-19) in China]. Zhonghua Liu Xing Bing Xue Za Zhi. 2020 Feb 10;41(2):145-151. doi: 10.3760/cma.j.issn.0254-6450.2020.02.003. Chinese. PMID 32064853
- [Result] Sockalingam S, Leung SE, Cassin SE. The Impact of Coronavirus Disease 2019 on Bariatric Surgery: Redefining Psychosocial Care. Obesity (Silver Spring). 2020 Jun;28(6):1010-1012. doi: 10.1002/oby.22836. PMID 32294297